CLINICAL TRIAL: NCT06433375
Title: Evaluation of the Efficacy of Growth Hormone, EndoSeal MTA Sealer, and Their Combination on Healing of Periapical Pathosis(Non-Surgical Approach)
Brief Title: Evaluation of the Efficacy of Growth Hormone, EndoSeal MTA Sealer, and Their Combination on Healing of Periapical Pathosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Zakaria Abd El Aziz, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27/4/2023
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Growth Hormone; EndoSeal MTA; Periapical Pathosis
Keywords: Periapical Pathosis; Growth Hormone; EndoSeal MTA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth hormone group (Experimental): Teeth undergo Growth Hormone application before obturation using EndoSeal MTA sealer
  Interventions: Procedure: Growth hormone application
- Control group (Experimental): Teeth undergo conventional root canal obturation using EndoSeal MTA sealer without any additional intervention
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Growth hormone application — Growth hormone application during non-surgical root canal treatment
  Arms: Growth hormone group
Procedure: Root canal treatment — Teeth undergo conventional root canal treatment without any additional intervention
  Arms: Control group

SUMMARY:
This study aimed to evaluate the effect of growth hormone, EndoSeal MTA sealer, and their combination on Healing of Periapical Pathosis.

DETAILED DESCRIPTION:
Out of 100 healthy male patients aged 18 to 40 years, 32 were selected from outpatients attending the Endodontic Clinic of the Faculty of Dental Medicine, Al-Azhar University, Cairo, Egypt, to be included in this study. The selected patients have no medical contraindications for oral surgical procedures (Scores 1-2) according to the classification of the American Society of Anesthesiologists (ASA)(8). Single-rooted permanent teeth were selected according to specific inclusion criteria based on preoperative assessment of the patients.

ELIGIBILITY:
Inclusion Criteria:- Necrotic teeth with apical periodontitis.

* Teeth presented with normal pocket depth ranges from 1 to 3mm, up to grade II tooth mobility.
* Teeth with mature apices, root canal curvature between (0-10º) according to Schneider(9) and radii of curvature between 2 to 5 mm according to Pruett would be included in the study(10).
* Teeth with estimated working length of 20mm(±2mm) from the incisal edge as a reference point provided that the crown/root ratio was not compromised.
* Non-critical sized periapical lesion related only to one tooth of a 2 to 4mm diameter and score 3 when evaluated using the Cone Beam Computed Tomography Periapical Index Score (CBCTPAI)(11) , Table (1) presents the scoring scale of CBCT-PAI.
* Teeth located in anatomic areas in which enucleation of the periapical tissues may jeopardize nearby structures, such as the incisive foramen or nasal cavity should be at least 2 mm away from these structures.

Exclusion Criteria:

* Necrotic teeth with related periapical swelling or sinus tract.
* Teeth with previous root canal fillings and /or indirect coronal restoration.
* Teeth with abnormal root canal anatomy.
* Non-restorable teeth due to insufficient coronal tooth structure.
* Teeth with periodontal disease.
* Teeth with grade III mobility.
* Teeth with clinical evidence of a missing buccal bony plate over the periapical defect.
* Traumatized teeth with suspected root cracks, fractures, intrusive and extrusive injuries, previously avulsed or lateral luxation injuries.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Post operative CBCT scan | 6 months
  Evaluation of non surgical root canal tratment healing according to CBCTPAI
Post operative CBCT scan | 12 months
  Evaluation of non surgical root canal tratment healing according to CBCTPAI

SECONDARY OUTCOMES:
Post operative pain assesment | 6 hours
  The postoperative pain assessment was done after obturation, using the modified verbal descriptor scale (VDS) as follow The VDS consist of a scoring system translated into an Arabic, describes a list of adjectives describing the different level of pain including, no pain (score 0 -1), mild pain (score 2-3), moderate pain (score 4 -5), strong pain (score 6 - 7), severe pain (score 8 - 9), worst pain (score 10).
Post operative pain assesment | 24 hours
  The postoperative pain assessment was done after obturation, using the modified verbal descriptor scale (VDS) as follow The VDS consist of a scoring system translated into an Arabic, describes a list of adjectives describing the different level of pain including, no pain (score 0 -1), mild pain (score 2-3), moderate pain (score 4 -5), strong pain (score 6 - 7), severe pain (score 8 - 9), worst pain (score 10).
Post operative pain assesment | 48 hours
  The postoperative pain assessment was done after obturation, using the modified verbal descriptor scale (VDS) as follow The VDS consist of a scoring system translated into an Arabic, describes a list of adjectives describing the different level of pain including, no pain (score 0 -1), mild pain (score 2-3), moderate pain (score 4 -5), strong pain (score 6 - 7), severe pain (score 8 - 9), worst pain (score 10).
Post operative pain assesment | 72 hours
  The postoperative pain assessment was done after obturation, using the modified verbal descriptor scale (VDS) as follow The VDS consist of a scoring system translated into an Arabic, describes a list of adjectives describing the different level of pain including, no pain (score 0 -1), mild pain (score 2-3), moderate pain (score 4 -5), strong pain (score 6 - 7), severe pain (score 8 - 9), worst pain (score 10).
Post operative pain assesment | 1 week
  The postoperative pain assessment was done after obturation, using the modified verbal descriptor scale (VDS) as follow The VDS consist of a scoring system translated into an Arabic, describes a list of adjectives describing the different level of pain including, no pain (score 0 -1), mild pain (score 2-3), moderate pain (score 4 -5), strong pain (score 6 - 7), severe pain (score 8 - 9), worst pain (score 10).

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Nasr City, Egypt